CLINICAL TRIAL: NCT01158040
Title: Intrapartum Maternal Glycemic Control Using Insulin Pump Versus Insulin Drip Cohort Retrospective and Prospective Observational Trial
Brief Title: Intrapartum Maternal Glycemic Control Using Insulin Pump Versus Insulin Drip - Cohort Observational Trial
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Hagit Shani MD, Sheba Medical Center
Other Study IDs: SHEBA-10-8014-HS-CTIL
Record Dates: First submitted 2010-07-04; First posted 2010-07-08 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Pregestational Diabetes
Keywords: Maternal intrapartum glycemic control; Pregestational diabetes

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Insulin pump: Women suffering from pregestational diabetes mellitus and being treated with insulin pump during pregnancy and delivery
- IV insulin: Women suffering from pregestational diabetes mellitus and being treated with insulin sub-cutan (SC) during pregnancy and IV insulin during delivery
- Healthy: Healthy women accepted for delivery in our institute

SUMMARY:
The purpose of this study is to compare intrapartum glycemic control using insulin pump versus intravenous (IV) insulin administration.

DETAILED DESCRIPTION:
Intrapartum maternal glycemic control in women suffering from pregestational diabetes mellitus type 1 will be evaluated and compared in the 3 study groups. Maternal and neonatal capillary blood glucose will be measured. All women suffering from diabetes mellitus and all neonates to hyperglycemic mothers are being tested for their blood glucose in our institute. Measurements' data will be collected. The primary outcome of the study is the number of neonatal hypoglycemic events (neonatal blood glucose < 40mg/dL). All women participating in the study will be treated according to the standard accepted protocol for "the treatment of pregestational diabetes during labor" in our institute. The research will not include new treatments or equipment.

The study is a cohort prospective and retrospective observational study in the tertiary center - Sheba medical center.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women suffering from pregestational diabetes mellitus type-1,
* Women are being treated for a minimum of 3 months in the high risk pregnancy clinic in Sheba medical center
* Women are being treated with either insulin pump or SC insulin (basal-bolus)

Exclusion Criteria:

* Women not compliant to treatment
* Women not planning their delivery in our institute

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women suffering from pregestational diabetes mellitus type-1, and are being treated for a minimum of 3 months in the high risk pregnancy clinic in Sheba medical center.
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Neonatal hypoglycemia (neonatal capillary blood glucose lowers then 40 mg/dL) | Up to 2 hours postpartum
  All neonates to mothers who suffer from diabetes mellitus are being routinely tested for neonatal hypoglycemia in our department. Their capillary blood glucose level is being tested in the first 2 hours postpartum. Data will be gathered and compared in women being treated with insulin pump during labor versus women being treated with IV insulin

SECONDARY OUTCOMES:
Mean maternal blood glucose during labor | Over the course of delivery
  All women suffering from pregestational diabetes mellitus are being routinely tested for blood glucose levels during delivery in our department. Their capillary blood glucose level is being tested every 1 hour throughout the active phase of delivery. Mean maternal blood glucose during partum will be compared in women being treated with insulin pump during labor versus women being treated with IV insulin

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Sivan, MD. PROF, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Taylor R, Lee C, Kyne-Grzebalski D, Marshall SM, Davison JM. Clinical outcomes of pregnancy in women with type 1 diabetes(1). Obstet Gynecol. 2002 Apr;99(4):537-41. doi: 10.1016/s0029-7844(01)01790-2. PMID 12039106
- [Background] Lepercq J, Abbou H, Agostini C, Toubas F, Francoual C, Velho G, Dubois-Laforgue D, Timsit J. A standardized protocol to achieve normoglycaemia during labour and delivery in women with type 1 diabetes. Diabetes Metab. 2008 Feb;34(1):33-7. doi: 10.1016/j.diabet.2007.08.003. PMID 18069031
- [Background] Jovanovic L. Glucose and insulin requirements during labor and delivery: the case for normoglycemia in pregnancies complicated by diabetes. Endocr Pract. 2004 Mar-Apr;10 Suppl 2:40-5. doi: 10.4158/EP.10.S2.40. PMID 15251639
- [Background] Carron Brown S, Kyne-Grzebalski D, Mwangi B, Taylor R. Effect of management policy upon 120 Type 1 diabetic pregnancies: policy decisions in practice. Diabet Med. 1999 Jul;16(7):573-8. doi: 10.1046/j.1464-5491.1999.00124.x. PMID 10445833
- See also: ACOG Committee practice bulletins — http://www.ncbi.nlm.nih.gov/sites/pubmed